CLINICAL TRIAL: NCT06231576
Title: Digital Home-Based Prehabilitation Before Surgery
Acronym: dHOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23/08551
Record Dates: First submitted 2023-11-17; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cancer Colorectal; Frailty; Surgery
Keywords: Prehabilitation; Colorectal cancer; Frailty
MeSH Terms: conditions — Colonic Neoplasms; Frailty; Colorectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hospital (Experimental): Prehabilitation at the hospital, with guidance by a dedicated physiotherapist physically present.
  Interventions: Other: Prehabilitation
- Digital (Experimental): Prehabilitation at home, with guidance from a dedicated physiotherapist through a digital platform, realtime.
  Interventions: Other: Prehabilitation
- Control (No Intervention): Information about the general benefit of a healthy lifestyle at inclusion, thereafter no further follow-up prior to surgery.

INTERVENTIONS:
Other: Prehabilitation — * Nutritional optimization: A nutritionist will perform a structured interview, comprehensive nutrition assessment, and provide personalized dietary advice. The main goal is to ensure optimal protein intake to support exercise-induced anabolism. A daily protein intake of 1.2-2.0 g/kg will meet needs as outlined in surgical nutrition guidelines.
  * Exercise: Based on current guidelines and instructed by a dedicated physiotherapist, for 1 hour per day preoperatively to increase muscle strength, aerobic capacity and physical endurance. Intensity will be based on the rate of perceived exertion using the Borg scale, a 15-graded scale ranging from very light to very hard. Resistance exercises will target upper/lower body, and abdominal muscles.
  * Psychological coaching and support: Performed as one interview during inclusion, followed by weekly phone calls by a study nurse coordinator during the preoperative intervention.
  Arms: Digital; Hospital

SUMMARY:
This clinical trial compares two different prehabilitation programs, with no organized prehabilitation, prior to major colorectal cancer surgery. The prehabilitation programs include intensive and coached physical exercise and optimized nutritional intake coupled with smoking cessation, physiological support and correction of poly-pharmacy.

DETAILED DESCRIPTION:
Patients are randomized to either a digital home-based program, a physical hospital-based program or no-organized prehabilitation. The eligible patients are anyone scheduled for colorectal cancer surgery who are fluent in Norwegian able to consent and to understand questionnaires. The main question the study aims to answer is whether a digital home-based program is non-inferior to a hospital-based program in terms of improved physical capacity and maintenance of life-quality. In addition, blood samples will be drawn at three time points, at inclusion, after intervention (prior to surgery) and 6 weeks after surgery to analyze and search for biomarkers reflecting patients' individual surgical risk profile and response to prehabilitation. Participants randomized to intervention, will be given psychological coaching and support, individualized nutritionist counselling, coached, structured and repeated 60 minutes daily exercises for three weeks prior to surgery. The control group will receive no organized prehabilitation in the period of time between diagnose and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned for major gastrointestinal cancer surgery
* Fluent in Norwegian and able to consent and to understand questionnaires

Exclusion Criteria:

* Inability to walk for six minutes or to rise independently from a chair
* Inability to comprehend exercise program or to comply with written and oral instructions
* Presence of a cardio-pulmonary condition that precludes exercise
* Living in very remote areas making a hospital-based intervention group impossible to implement
* Being without a permanent address
* Admittance to a hospital facility for > 50% of the time from diagnosis to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
6MWT | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  Distance (in meters) walked in 6 minutes

SECONDARY OUTCOMES:
EuroQol Group Questionnaire 5D (EQ-5D) | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  EQ-5D is a standardized measure of health-related quality of life with 5 dimensions, each dimension represented by a value 1-5 where higher value represents worse outcome.
European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Generic Short Patient Experiences Questionnaire (GS-PEQ) | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  GS-PEQ is a questionnaire for collecting data about user experiences across different types of services. The questionnaire has 12 questions ranging from 1-5; a higher score represents a higher ("better") experience.
Mortality | 3 months after surgery
  90-day mortality
Complications | 3 months after surgery
  Comprehensive Complication Index (CCI) reflects the gravity of the overall complication burden on the patient on a scale from 0 (no complication) to 100 (death)
Need of additional health care support | 4-6 weeks after surgery
  Use of health care support from the municipality, nursing homes etc
Aggregated length-of-stay (aLoS) | 4-6 weeks after surgery
  Total time in hospital (from surgery and any readmittance) within 30-days from surgery
Cost-effectiveness | 3 months after surgery
  An estimation of the resources used on the prehabilitation program will be compared to resources saved by shorter aLoS, less use of nursing home facilities and less need of community healthcare services

OTHER OUTCOMES:
DNA methylation | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  Blood samples for DNA methylation profiling will be implemented in a machine learning algorithm to search for biomarkers reliably reflecting frailty and effect of prehabilitation.
RNA methylation | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  Blood samples for RNA methylation profiling will be implemented in a machine learning algorithm to search for biomarkers reliably reflecting frailty and effect of prehabilitation.
Metabolome | At inclusion, prior to intervention. After intervention, prior to surgery. 4-6 weeks after surgery
  Blood samples for metabolome profiling will be implemented in a machine learning algorithm to search for biomarkers reliably reflecting frailty and effect of prehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Rune Ougland, MD PhD, Principal Investigator — Vestre Viken, Bærum Hospital, Norway

IPD SHARING:
Plan to Share IPD: Yes
Protocol and SAP will be published together with results from the pilot study
Supporting Information: Study Protocol, SAP
Time Frame: By end of 2024
Access Criteria: Upon request

REFERENCES:
- [Derived] Kleve G, Santa CD, Kristiansen F, Tegnander M, Buch V, Hagemann CS, Helgheim M, Engene P, Pesonen H, Kleveland MK, Hverven GL, Nilsen TS, Vervaart MAM, Aanesen H, Uglane KT, Bjelland M, Zory R, Chorin F, Cardot-Ruffino V, Beltran EEM, Neuzillet C, Soerensen M, Jylhava J, Anzar I, Normand VA, Myrstad M, Klungland A, Nilsen HL, Ougland R. Digital home-based multimodal prehabilitation of colorectal cancer patients prior to surgery (the dHOPE study): a non-inferiority clinical trial protocol. Front Digit Health. 2025 Oct 8;7:1609678. doi: 10.3389/fdgth.2025.1609678. eCollection 2025. PMID 41132395

DOCUMENTS (1):
  • Study Protocol (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT06231576/Prot_000.pdf